CLINICAL TRIAL: NCT03998371
Title: Ultrasensitive Chromosomal Aneuploidy Detection (UCAD) in Urine Exfoliated Cells for Diagnosis of Urothelial Carcinoma in in Urine Exfoliated Cells
Brief Title: Application of UCAD for Diagnosing Urothelial Carcinoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Shuxiong Zeng, Principal Investigator, Changhai Hospital
Other Study IDs: CH-urology-bladder marker-002
Record Dates: First submitted 2019-06-19; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Urothelial Carcinoma; Diagnoses Disease; Chromosomal Abnormality; Urine Marking
Keywords: Urothelial Carcinoma; diagnosis; Chromosomal Aneuploidy Detection; marker; urine
MeSH Terms: conditions — Carcinoma, Transitional Cell; Chromosome Aberrations; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from Urine Exfoliated Cells will be analyzed by Ultrasensitive Chromosomal Aneuploidy Detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urothelial carcinoma group: Pre-surgery patients with urothelial carcinoma will be the experimental group to determine the sensitivity and specificity of UCAD analysis, the result will be compared with cytology and FISH.
  Interventions: Diagnostic Test: Low-coverage whole-genome sequencing of urine exfoliated cells
- Non-cancer participants group: Patients being treated for other diseases but without any tumor will provide a negative control to provide data for determining the sensitivity and specificity of UCAD analysis.
  Interventions: Diagnostic Test: Low-coverage whole-genome sequencing of urine exfoliated cells

INTERVENTIONS:
Diagnostic Test: Low-coverage whole-genome sequencing of urine exfoliated cells — The level of CIN The extracted DNA from morning urine will be analyzed by UCAD to determine the level of CIN.

SUMMARY:
Chromosomal instability (CIN) refers to ongoing chromosome segregation errors throughout consecutive cell divisions. CIN is a hallmark of human cancer, and it is associated with poor prognosis, metastasis, and therapeutic resistance. Analyzing CIN of the DNA extracted from urothelial cells in urine samples seems a promising method for diagnosing, monitoring, and predicting the prognosis of bladder cancer patients. CIN can be assessed using experimental techniques such as bulk DNA sequencing, fluorescence in situ hybridization (FISH), or conventional karyotyping. However, these techniques are either time-consuming or non-specific. We here intend to study whether a new method named Ultrasensitive Chromosomal Aneuploidy Detection (UCAD), which is based on low-coverage whole-genome sequencing, can be used to analyze CIN thus help diagnosing and treating bladder cancer patients.

DETAILED DESCRIPTION:
CIN results from errors in chromosome segregation during mitosis, leading to structural and numerical chromosomal abnormalities. It will generate genomic heterogeneity that acts as a substrate for natural selection. Furthermore, it is proved that tumors with aneuploidies and polyploidy resulting from whole-genome doubling are related with metastasis, treatment resistance, and decreased overall survival. It is estimated that 60%-80% of human tumors exhibit chromosomal abnormalities suggestive of CIN. CIN positively correlates with tumor stage and is enriched in relapsed as well as metastatic tumor specimens. Due to the ubiquity of CIN in cancer cells, it is a potentially non-invasive way to detect CIN in the urothelial cells from the urine sample for diagnosing and monitoring bladder cancer patients. UCAD is a new method to detecting CIN in the DNA sample from patients, including extracting DNA from urine, analyzing DNA by low-coverage whole-genome sequencing, processing the data by bio-information techniques, and finally optimizing the management of bladder cancer patients.

The investigators intended to conduct a prospective study by analyzing urine samples from bladder cancer patients and control groups that without any tumor in the urinary system or other organs to compare the specificity and sensitivity of UCAD test for diagnosing urothelial carcinoma to other modalities, such as urine cytology or fluorescence in situ hybridization (FISH).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with urothelial carcinoma and planned to undergo surgery.
* Participants without any tumor disease and willing to attend the study by providing morning urine.
* Male or female patients aged >= 18 years.
* Participants signed informed consent form.

Exclusion Criteria:

* Age under 18 years
* Individuals unwilling to sign the consent form or unwilling to provide morning urine for test or unwilling to provide the medical record.
* Individuals unwilling to participate in this trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with urothelial carcinoma or participants in control group in Changhai Hospital from May 2019 till the end of this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of urinalysis by UCAD analysis | Up to 1 years
  Number of patients "declared positive" with the UCAD test among the patients suffered from urothelial carcinoma.
Specificity of urinalysis by UCAD analysis | Through study completion, an average of 12 months
  Number of patients "declared negative" with the UCAD test among the patients without cancer.

SECONDARY OUTCOMES:
Comparison of the sensitivity of the UCAD analysis versus urine cytology | Up to 1 years
  Number of patients "declared positive" with the UCAD analysis versus patients "declared positive" with the urine cytology.
Comparison of the specificity of the UCAD analysis versus urine cytology | Up to 1 years
  Number of patients "declared negative" with the UCAD analysis versus patients " declared negative " with the urine cytology.

OTHER OUTCOMES:
Identification of the correlation between the level of CIN and the grade of the tumor sample | Up to 1 years
  Level of CIN in the urine sample compared with the grade of the tumor confirmed by histopathologic examination
Identification of the correlation between the level of CIN and the stage of the tumor sample | Up to 1 years
  Level of CIN in the urine sample compared with the stage of the tumor confirmed by histopathologic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Chuangliang Xu, M.D., Ph.D, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We will try to protect the information of the included participants

REFERENCES:
- [Background] Wadhwa N, Mathew BB, Jatawa SK, Tiwari A. Genetic instability in urinary bladder cancer: An evolving hallmark. J Postgrad Med. 2013 Oct-Dec;59(4):284-8. doi: 10.4103/0022-3859.123156. PMID 24346386
- [Background] Bakhoum SF, Ngo B, Laughney AM, Cavallo JA, Murphy CJ, Ly P, Shah P, Sriram RK, Watkins TBK, Taunk NK, Duran M, Pauli C, Shaw C, Chadalavada K, Rajasekhar VK, Genovese G, Venkatesan S, Birkbak NJ, McGranahan N, Lundquist M, LaPlant Q, Healey JH, Elemento O, Chung CH, Lee NY, Imielenski M, Nanjangud G, Pe'er D, Cleveland DW, Powell SN, Lammerding J, Swanton C, Cantley LC. Chromosomal instability drives metastasis through a cytosolic DNA response. Nature. 2018 Jan 25;553(7689):467-472. doi: 10.1038/nature25432. Epub 2018 Jan 17. PMID 29342134
- [Background] Liu H, He W, Wang B, Xu K, Han J, Zheng J, Ren J, Shao L, Bo S, Lu S, Lin T, Huang J. MALBAC-based chromosomal imbalance analysis: a novel technique enabling effective non-invasive diagnosis and monitoring of bladder cancer. BMC Cancer. 2018 Jun 15;18(1):659. doi: 10.1186/s12885-018-4571-7. PMID 29907142
- [Background] Hieronymus H, Murali R, Tin A, Yadav K, Abida W, Moller H, Berney D, Scher H, Carver B, Scardino P, Schultz N, Taylor B, Vickers A, Cuzick J, Sawyers CL. Tumor copy number alteration burden is a pan-cancer prognostic factor associated with recurrence and death. Elife. 2018 Sep 4;7:e37294. doi: 10.7554/eLife.37294. PMID 30178746
- [Derived] Zeng S, Ying Y, Xing N, Wang B, Qian Z, Zhou Z, Zhang Z, Xu W, Wang H, Dai L, Gao L, Zhou T, Ji J, Xu C. Noninvasive Detection of Urothelial Carcinoma by Cost-effective Low-coverage Whole-genome Sequencing from Urine-Exfoliated Cell DNA. Clin Cancer Res. 2020 Nov 1;26(21):5646-5654. doi: 10.1158/1078-0432.CCR-20-0401. Epub 2020 Oct 9. PMID 33037018